CLINICAL TRIAL: NCT07030231
Title: Utilización de la Radioterapia IntraOperatoria en la Neoplasia de MAma
Brief Title: Use of Intraoperative Radiotherapy in Breast Cancer
Acronym: RIOMA
Status: Enrolling by invitation | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Manuel Algara, Principal Investigator, Parc de Salut Mar
Other Study IDs: SESPM-19-1
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: Breast Cancer; Intraoperative radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Intraoperative — Intraoperative radiotherapy with any device after conservative surgery in early breast cancer

SUMMARY:
The Utility of Intraoperative Radiotherapy in Breast Cancer (RIOMA) is an observational project to understand the use and outcomes of intraoperative radiotherapy in patients with breast cancer under conditions of clinical use (not clinical trials). Intraoperative radiotherapy (IORT) is a technique that began to be used years ago, transferring the patient from the operating room to the radiotherapy suite. This technique therefore fell into disuse. The emergence of miniaturized linear accelerators has led to a resurgence of IORT, especially as part of conservative treatment in patients with breast cancer, both as a booster or as a sole treatment (partial breast irradiation).

This project is based on an online platform. Each participating center will be assigned access codes on the website to access and complete the coded clinical data for each patient treated with intraoperative radiotherapy. Data on tumor characteristics, the type of intraoperative radiotherapy, follow-up, complications, and cosmetic outcomes are included.

Primary objective:

To understand the characteristics of patients treated with intraoperative radiotherapy under routine clinical practice conditions.

DETAILED DESCRIPTION:
The project is based on structured data collection in an electronic data collection notebook (using the OpenclinicaTM standard), relating to the care provided according to standard clinical practice in the Radiation Oncology, Gynecology and Surgery departments of the participating centers in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer who are candidates for intraoperative irradiation exclusively
* Patients with breast cancer who are candidates for intraoperative irradiation combined with external beam irradiation
* Patients with recurrence of breast cancer who are candidates for intraoperative irradiation
* Have read the information sheet and signed the informed consent form -

Exclusion Criteria:

* Patient's that express wish not to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early breast cancer who are candidates for intraoperative radiotherapy, such as exclusive partial irradiation, anticipated boosting, or salvage after a second conservative surgery.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2030-04-01 (Estimated); Study Completion 2031-04-01 (Estimated)

PRIMARY OUTCOMES:
Characteristics of patients treated with intraoperative radiotherapy according to the conditions of standard clinical practice, | From enrollement to the end of recruitment at 10 years
  To evaluate the characteristics of patients treated with intraoperative radiotherapy according to the conditions of standard clinical practice, retrospectively from the beginning of the implementation of the technique and prospectively from the launch of this registry.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Barcelona, Spain